CLINICAL TRIAL: NCT04004819
Title: Rituximab Therapy for the Patients With HTLV-1-associated Myelopathy
Brief Title: Rituximab for HTLV-1-associated Myelopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Wan-Jin Chen, Neurology department, First Affiliated Hospital of Fujian Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRCTA,ECFAHOFFMU[2019]142
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: HTLV-1-associated Myelopathy
MeSH Terms: conditions — Paraparesis, Tropical Spastic | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: Experimental: Rituximab group Drug: Rituximab will be administered as 100 mg IV, once per week for 3 consecutive weeks. Continued dosage was dependent on the percentage of circulating CD19 B-cell counts from patients . Whenever it reached 1% of total lymphocyte population, rituximab 100 mg was reinfused
  Placebo Comparator: Control group Patients will receive usual care and drug use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab group (Experimental): Rituximab will be administered as 100 mg IV, once per week for 3 consecutive weeks. Continued dosage was dependent on the percentage of circulating CD19 B-cell counts from patients . Whenever it reached 1% of total lymphocyte population, rituximab 100 mg was reinfused
  Interventions: Drug: Rituximab
- Control group (No Intervention): Patients will receive usual care and drug use.

INTERVENTIONS:
Drug: Rituximab — A lower dosage of rituximab for HTLV-1-associated myelopathy
  Arms: Rituximab group

SUMMARY:
Neuroprotective or anti-inflammatory strategies are invaluable in HTLV-1-associated myelopathy due to its rapid progression. We evaluated the efficacy of rituximab in patients with HTLV-1-associated myelopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Patients HTLV-1-associated myelopathy (tropical spastic paraparesis)

Exclusion Criteria:

* Anticipated survival of at least 3 years
* Inability to undergo neuroimaging with Magnetic Resonance
* Clinically significant hepatic disease as demonstrated by history, clinical exam (ascites, varices), or laboratory findings (LFTs >2x normal, coagulopathy as described)
* Comorbid conditions likely to complicate therapy including but not limited to the following: a history of New York Heart Association class II, III, or IV Congestive Heart Failure; end-stage acquired immune deficiency syndrome
* Pregnancy
* Malignancy (history of or active)
* Concomitant use with antineoplastic, immunosuppressive or immune modulating therapies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
The improvement of pyramidal or bowel-bladder function score in EDSS during 12 month treatment | up to 360 days
  EDSS include the evaluated on visual, brainstem, pyramidal, cerebellar, sensory, bowel-bladder and cerebral functions

SECONDARY OUTCOMES:
Change in immunology function | up to 360 days
  Use the flow cytometry to measure the change at baseline, 90,180, 360 days after drug use

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology ,First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Lv A, Fang Y, Lin X, Chen J, Song H, Wang N, Chen WJ, Fu Y, Li R, Lin Y. B-cell depletion limits HTLV-1-infected T-cell expansion and ameliorate HTLV-1-associated myelopathy. Ann Clin Transl Neurol. 2024 Oct;11(10):2756-2768. doi: 10.1002/acn3.52190. Epub 2024 Aug 26. PMID 39186315